CLINICAL TRIAL: NCT06582888
Title: Advancing VR-based Attentional Bias as a Biomarker for Tobacco Use Disorder
Acronym: VR
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kelly Courtney, Assistant Adjunct Professor, Psychiatry, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: R01DA058665 (NIH); R01DA058665 (NIH)
Record Dates: First submitted 2024-08-21; First posted 2024-09-03 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Nicotine Addiction; Craving
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Varenicline

STUDY DESIGN:
Intervention Model Description: The proposed project will include enrollment of 200 daily tobacco cigarette users, ages 22+, from the San Diego community. Participants will be assessed on the VR Nicotine Cue Exposure paradigm then randomized (stratified on age and sex) to receive varenicline (target dose 1mg twice daily) or placebo (n per group=100; total N=200). Following eight days of titration, participants will be assessed again on the VR Nicotine Cue Exposure paradigm. They will then be followed via mobile assessments for eight days on target dose of varenicline, and 30-days post assessment by phone, to assess short-term nicotine use behaviors.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Varenicline (Experimental): Following the baseline assessment, participants randomized to receive varenicline will complete an 8-day titration period to achieve the target dose. Titration of varenicline will be as follows: 0.5 mg once daily for Days 1-3, 0.5 mg twice daily for Days 4-7, and 1 mg twice daily on Day 8. Participants then return to the lab on Day 9 (or Days 10, 11 if necessary) for testing at the target dosage (1 mg twice daily) and continue at that dose for eight additional days (Days 10-17) for mobile monitoring.
  Interventions: Drug: Varenicline Tartrate
- Placebo (Placebo Comparator): Following the baseline assessment, participants randomized to receive placebo pill will follow the same dosing schedule as the active arm. They will return to the lab on Day 9 (or Days 10, 11 if necessary) for testing and continue at that dosing schedule for eight additional days (Days 10-17) for mobile monitoring.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline Tartrate — varenicline (target dose 1mg twice daily)
  Other Names: Varenicline
  Arms: Varenicline
Drug: Placebo — matched placebo
  Arms: Placebo

SUMMARY:
The proposed project will include enrollment of 200 daily tobacco cigarette users, ages 22+, from the San Diego community. Participants will be assessed on the VR Nicotine Cue Exposure paradigm then randomized (stratified on age and sex) to receive varenicline (target dose 1mg twice daily) or placebo (n per group=100; total N=200). Following eight days of titration, participants will be assessed again on the VR Nicotine Cue Exposure paradigm. They will then be followed via mobile assessments for eight days on target dose of varenicline, and 30-days post assessment by phone, to assess short-term nicotine use behaviors.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Persons, aged 22+
4. Ability to take oral medication and be willing to adhere to the dosing regimen
5. For participants able to become pregnant: use of highly effective contraception during study enrollment
6. Current daily tobacco use (use on 7 days per week, on average, ≥5 cigarettes per day, in the previous 3 months)
7. Tobacco use history ≥3 years
8. Endorsement of past week nicotine craving

Exclusion Criteria:

1. Contraindications/conditions with special precautions for varenicline treatment (i.e., history of serious hypersensitivity or skin reactions to varenicline, history of severe renal impairment, seizures, severe cardiovascular disease, chronic or severe nausea, Stevens-Johnson syndrome, erythema multiforme, pregnancy or nursing)
2. Medical or psychiatric history affecting brain development (i.e., history and/or treatment of neurologic disorders, severe head trauma with loss of consciousness >2 minutes, or current severe Diagnostic and Statistical Manual 5th edition (DSM-5) psychiatric disorders other than tobacco use disorders)
3. Current suicidal ideation or history of suicide attempt or self-mutilatory acts in the past 12 months
4. Other recreational drug use in the past 30 days (besides alcohol and cannabis) verified by oral and urine fluid toxicology
5. Visual/vestibular problems that may make task completion difficult (i.e., motion sickness, difficulty balancing, blindness)
6. Treatment seeking for tobacco use disorder/intent to quit within 30 days

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2028-08-15 (Estimated); Study Completion 2028-08-15 (Estimated)

PRIMARY OUTCOMES:
Change in Virtual Reality Attentional Bias (VR-AB) pre- and post-treatment | during each in-person session, at baseline and on average 8 days post baseline assessment
  Eye gaze fixation time to active versus neutral cues from the "NTP Cue VR Paradigm"
Nicotine craving | during each in-person session, at baseline and on average 8 days post baseline assessment
  Assessed via the Tobacco Craving Questionnaire - Short-Form
Nicotine craving | through study completion, an average of 30 days
  Assessed via visual analogue scales (VR paradigm and mobile surveys)
Nicotine use episodes | during each in-person session, at baseline and on average 8 days post baseline assessment
  Assessed via the Timeline Followback
Nicotine use episodes | through study completion, an average of 30 days
  Assessed via participant fill-in on mobile surveys

CONTACTS AND LOCATIONS:
Locations (1):
- University California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Psychophysiology, mental health, and substance use de-identified data listed above sufficient in quality to validate and replicate the research findings described in the aims will be deposited to the National Addiction & HIV Data Archive Program (NAHDAP) repository. For specific variables where small sample sizes may allow for easy re-identification of research participants, only summarized data will be made available.
Supporting Information: ICF, Analytic Code
Time Frame: Data will become available 2025-2028
Access Criteria: Standard procedures of the NAHDAP will be followed for determining the best level of access (public or restricted) based on review of disclosure risk by ICPSR.
URL: https://www.icpsr.umich.edu/web/pages/NAHDAP/index.html